CLINICAL TRIAL: NCT07385027
Title: LOVEH: Linked Outcomes in Various EEG-Hyperscanning Setups
Brief Title: Linked Outcomes in Various EEG-Hyperscanning Setups
Acronym: LOVEH
Status: Recruiting | Type: Observational
Sponsor: Spaulding Rehabilitation Hospital (Other)
Collaborators: Université de Montréal (Other); Brigham and Women's Hospital (Other); Emerald Gate Charitable Trust (Unknown)
Responsible Party: Principal Investigator, Alessandra Anzolin, Instructor, Spaulding Rehabilitation Hospital
Other Study IDs: 2025P000921
Record Dates: First submitted 2026-01-22; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Brain to Brain Communication
Keywords: Hyperscanning; EEG; Brain to Brain Communication; Healthy Control

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Romantic Pair: Two people involved in a romantic relationship for longer than 1 year.
  This is a cross-sectional study in which every subject will complete the experiment in both conditions, once with their romantic pair, and once with a randomly assigned stranger. Therefore, participants will complete one EEG with their romantic pair, and one EEG with a stranger. The order of the EEG scans and the cross-over will be randomized.
- Stranger Pair: Two people who have never seen each other before the EEG visit.
  This is a cross-sectional study in which every subject will complete the experiment in both conditions, once with their romantic pair, and once with a randomly assigned stranger. Therefore, participants will complete one EEG with their romantic pair, and one EEG with a stranger. The order of the EEG scans and the cross-over will be randomized.

SUMMARY:
The goal of this observational study is to investigate how brains of healthy controls respond when they interact with their romantic partner compared to when they interact with a stranger. The main goals are:

* Explore how two people's brains interact with each other by recording brain activity at the same time (a method called "hyperscanning") using electroencephalography (EEG). Using hyperscanning, this study will compare brain-to-brain communication in romantic couples versus strangers, both when they are together in person and when they are interacting remotely.
* Test a computational model that will help explain how this brain-to-brain communication works, using real data from the brain activity EEG recordings.
* Explore whether factors such as age, gender, how aware people are of their own body sensations, and their level of attachment influence brain-to-brain communication.

Researchers will compare brain-to-brain communication in romantic couples versus strangers, both when they are together in person and when they are interacting remotely to see which factors effect brain-to-brain communication.

Enrolled participants will:

* Complete a consent visit with their romantic partner where they will sign a consent form and have their pain sensitivity assessed.
* Fill out sets of questionnaires assessing their romantic relationship, their personality, and other traits.
* Complete two EEG scans, one with their romantic partner and one with a stranger. At both scans they will conduct a pain task, a communication task, and a light stimulation task.

DETAILED DESCRIPTION:
Twenty romantic pair dyads will be recruited for this study, for a total of 40 participants. Male and female participants, aged 20-60, will be recruited using Mass General Brigham (MGB) approved recruitment methods, specifically Rally. Subject recruitment will be conducted by primary investigators and study staff. Interested patients who filled out the Rally form will be sent a screening survey in RedCap, a secure online data capture system approved by MGB Human Research Committee, via a public link. Patients will be offered the alternative of a telephone screening if they are uncomfortable with this method. After successful RedCap or telephone screening, romantic pairs will be invited to our laboratory to undergo consent. At the consent visit, romantic pairs will sign the consent form, fill out baseline questionnaires, and assess their pain sensitivity using cuff pressure. Upon completing the consent visit, patients will proceed to a baseline EEG scan with either their romantic partner or a stranger, the order will be randomized. Each member of the romantic pair will be randomized to a different stranger. The participants will then complete a second EEG scan with either their romantic pair or a stranger, depending on which person they were randomized to during their first EEG scan.

At both of the EEG scans, participants will complete a variety of tasks both face-to-face and in remote settings. The two participants will be seated face to face with the EEG caps on for the face-to-face portion of the EEG experiment, and they will be in separate rooms for the remote part of the experiment. First, an EEG cap will be placed on the head of the both the participants and the signal quality will be assessed.

The participants will then start by completing 3 minutes of eyes open and 3 minutes of eyes closed rest. This will be repeated for both face-to-face and remote settings. Participants will additionally complete an intermittent light stimulation task (ILS) where a series of photic flashes delivered by a strobe light simulation on a high frame rate monitor placed 30cm from the participant's nose is presented to the participants with eyes closed. This task will be done both face-to-face as well as remotely. The ILS task includes three conditions, one where both participants receive light stimulation simultaneously, another two where each participant will receive light stimulation while the other participant receives no light stimulation. This task measures brain to brain communication in a controlled context and takes about 6 minutes.

Participants will additionally complete a communication task in which participants are asked to make a positive wish and send warm thoughts or love to the respective other (non-verbal phase) and to say why they made this wish (verbal phase). This task will be done both face-to-face as well as remotely. In the face-to-face setting, both participants are asked to sit still and relax during eye contact. The participants are instructed to "Make a wish for the other person and tell them what you wished for them and why" (verbal phase). Then, participants are asked to focus their attention on each other and send warm thoughts or love to the respective other (non-verbal phase). In the remote setting, both participants are asked to sit still and relax. One participant will be designated as the sender and will be instructed to "Think of the person in the other room and then make a wish for them. When you've made the wish, say it out loud and describe why you wish them what you wished".

Participants will additionally complete a cuff pain task. A blood pressure cuff device will be place on one of the participant's left leg and will be used to deliver moderately painful stimulations, calibrated at the consent visit. After each painful stimulation, the subject wearing the cuff will be asked to rate the pain they felt on a scale from 0-100 where 0 is no pain and 100 is the most intense pain imaginable. Simultaneously, the other participant will rate the level of pain they believe their experimental partner felt on the same 0-100 scale. The participants will then repeat the task with switched roles and participant 2 will be receiving moderate painful stimulations. This cuff task will be performed both in-person and remotely to assess the difference in brain to brain communication associated with empathy for pain and pain relief.

Lastly, patients will each complete an interoceptive awareness task - a task assessing the extent to which participants are aware of their own body sensations. The participants are instructed to alternate between focusing on their heartbeat/breathing (interoception) and visual/auditory stimuli (exteroception). After each trial, they are asked to rate the intensity of their body sensation from "No Sensation" to "Extremely Strong".

At various points throughout the EEG scan, participants will be administered questionnaires to assess their romantic relationship, their personality, and other traits.

The duration for each visit in this study will be approximately one hour for the consent visit and 2.5 hours per imaging visit. Therefore, each patient will spend a total of ~6 hours in the study.

A record will be created for each research subject, labeled by their subject ID using the software RedCap. It is a secure online data capture system which allows us to store and manage surveys and a database containing the answers to our questionnaires, notes on visits, and dates of the visits. All study visits will take place at Spaulding Rehabilitation Hospital (SRH).

ELIGIBILITY:
Inclusion Criteria

1. Healthy volunteers in a romantic partnership for at least 6 months.
2. 20-60 years of age
3. Ability to fully understand and consent to study procedures.
4. Fluent in English
5. Are on stable doses of medication for 30 days prior to entering the study and agree not to change medications or dosages during the trial.

Exclusion Criteria:

1. Presence of any contraindications to EEG scanning.
2. Illicit drug or opioid use.
3. Epilepsy, seizures provoked by lights or a prior history of seizures.
4. Presence of any illness that is judged to interfere with the trial. For example: severe psychiatric disorders according to the DSM-IV manual.
5. Current chronic pain conditions.
6. Unwillingness to be audio recorded.
7. Unwillingness to receive brief experimental pain on the lower left leg.
8. Unwillingness to withhold from consuming marijuana 48 hours prior to scans.
9. Unwillingness to withhold from consuming nicotine 4 hours prior to scans.
10. Any impairment, activity, or situation that in the judgment of the Study Coordinator or Principal Investigator would prevent satisfactory completion of the study protocol.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Twenty healthy control romantic pair dyads will be recruited for this study, for a total of 40 participants. Male and female participants, aged 20-60, will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Inter-Brain Connectivity (IBC) | 1 year
  Brain to brain connectivity (or IBC) estimated on EEG-hyperscan data acquired simultaneously from two people (either romantic partners or strangers). The investigators hypothesize that IBC (density of connections):
  * will be modulated by the level of attachment (factor 1) regardless of subjects proximity (same room versus separate rooms, factor 2).
  * will be stronger during communication task and empathy for pain compared to resting state.
  * will be affected by demographical factors including age, sex, and race.

SECONDARY OUTCOMES:
Heart-beat Evoked Potentials (HEP) during Interoception Task | 1 year.
  The ability to process internal-body sensations (interoception awareness) can be assessed by brain-heart interaction measures such as the brain potential generated in the brain after each heartbeat (HEP). The investigators hypothesize that different levels of interoception awareness measured by validated questionnaires (MAIA):
  * will modulate HEP during interoception task
  * will correlate with measures of inter-brain connectivty.

OTHER OUTCOMES:
Autonomic concordance. | 1 year
  Autonomic concordance between two subjects will be assessed during face-to-face hyperscanning experiments. Expected Research Outcomes:
  * Identify increased autonomic concordance during the communication task compared to resting state.
  * Identify a significant effect of the factors age, sex, level of attachment.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandra Anzolin, PhD, Principal Investigator — Spaulding Rehabilitation Hospital
Locations (1):
- Spaulding Rehabilitation Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Per IRB guidelines.